CLINICAL TRIAL: NCT00782964
Title: Assessment of Therapeutic Strategies in Unipolar Depression With Incomplete Response to a Antidepressant Treatment in Regular Clinical Practicing.
Brief Title: Antidepressant Incomplete Response Depression
Acronym: DRIA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Teresa Díez, PhD, Local MC Neuroscience Therapeutic Area Manager, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-NES-DUM-2007/4
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder; SSRI resistant depression; strategies in depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Outpatient with major depressive disorder, who has a change in pharmacological therapeutical plan after an incomplete response or intolerance to a treatment with an adequate dosage of an antidepressant (SSRI/NSRI) (20-40 mg fluoxetine, 75-225 mg venlafaxine or equivalent) for at least 6 weeks.

SUMMARY:
Observational, non-interventional, longitudinal, prospective,multicenter, open label (No treatment is involved). 3 assessment will be carried out . The 1st one will be on baseline, the 2sd one after a significant change in pharmacological treatment and 3rd one after a second significant change in pharmacological treatment. If there isn´t any significant change in therapeutic plan a control assessment will be carry out in week 10th and 24th. A significant treatment change is defined as a change in SSRI/SNRI, to add another SSRI/SNRI or a augmentation treatment added to SSRI/SNRI. The primary objective is to describe therapeutical strategies (antidepressant change, association with another antidepressant or association with another treatment) in the management of patients with MDD with incomplete response or intolerance to an antidepressant after a first or a second failure; and when the psychiatrist decide a change of strategy. Secondary objectives include: 1 - To describe the clinic profile of depressive patients with incomplete response or intolerance to an antidepressant after a first or a second failure; 2- To describe the profile of patients based on therapeutic strategies used and number of therapeutic strategies; 4- Evaluate the use of health resource due to lack of fast onset of action, and social cost (productivity, care givers…); 5 - To associate clinical variable with therapeutic action by psychiatrist.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written inform consent
* Diagnosed of Major Depressive Disorder based on DSM-IV-TR
* Outpatient who has a change in pharmacological therapeutic plan after an incomplete response or intolerance to a treatment with an adequate dosage of an antidepressant (SSRI/NSRI) 5
* Able to understand and to comply with requirements of the study

Exclusion Criteria:

* Mental retardation
* To have been recruited in a clinical trial in the last 4 weeks or to have planned the inclusion in a clinical trial during the follow-up of this study
* MDD secondary to substance abuse or somatic illness
* Actual depressive episode with <4 weeks or >12 months of length
* Current treatment with >1 SSRI/SRNI or previous treatment with >1 SSRI/SRNI, augmentation treatment with SSRI/SRNI, intravenous antidepressant treatment, TMS, ECT or MAO

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient with major depressive disorder, who has a change in pharmacological therapeutic plan after an incomplete response or intolerance to a treatment with an adecuate dosage of an antidepresant (SSRI/NSRI) (20-40 mg fluoxetine, 75-225 mg venlafaxine or equivalent) for at least 6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2008-10; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Profile of use of 3 group of strategies: 1 - Change to another antidepressive agent (Quetiapine, Lamotrigine, antidepressant…) 2- Association with another antidepressant 3- Association with any other treatment (antipsychotics, lithium…) | Baseline, after a significant change in treatment (or control visit after 10th week) and after a 2sd significant change in treatment (or control visit after 24th week).

SECONDARY OUTCOMES:
Clinical assessment | Baseline, after a significant change in treatment (or control visit after 10th week) and after a 2sd significant change in treatment (or control visit after 24th week).
Visits to nurse, psychiatrics: Hospitalization, social support: Productivity assessment | Baseline, after a significant change in treatment (or control visit after 10th week) and after a 2sd significant change in treatment (or control visit after 24th week).

CONTACTS AND LOCATIONS:
Locations (48):
- Spain (48):
  - Research Site, Albacete, Albacete
  - Research Site, Alcoy, Alicante
  - Research Site, Benidorm, Alicante
  - Research Site, Villajoyosa, Alicante
  - Research Site, Almería, Almeria
  - Research Site, Mérida, Badajoz
  - Research Site, Inca, Balearic Islands
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, El Hospitalet de Llobregat, Barcelona
  - Research Site, Martorell, Barcelona
  - Research Site, Vic, Barcelona
  - Research Site, Burgos, Burgos
  - Research Site, San Fernando, Cadiz
  - Research Site, Villamartín, Cadiz
  - Research Site, Santander, Cantabria
  - Research Site, Murcia, Caravaca
  - Research Site, Villarreal, Castellon
  - Research Site, Ceuta, Ceuta
  - Research Site, Córdoba, Cordoba
  - Research Site, Guadix, Granada
  - Research Site, Arrasate / Mondragón, Guipuzcoa
  - Research Site, Las Palmas de Gran Canaria, Las Palmas
  - Research Site, Lleida, Lerida
  - Research Site, Alcalá de Henares, Madrid
  - Research Site, Alcobendas, Madrid
  - Research Site, Colmenar Viejo, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, Torrejón de Ardoz, Madrid
  - Research Site, Málaga, Malaga
  - Research Site, Cartagena, Murcia
  - Research Site, Pamplona, Navarre
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Salamanca, Salamanca
  - Research Site, Seville, Sevilla
  - Research Site, Tarragona, Tarragona
  - Research Site, Valls, Tarragona
  - Research Site, La Cuesta de Arguijon, Tenerife
  - Research Site, Santa Cruz de Tenerife, Tenerife
  - Research Site, Talavera de la Reina, Toledo
  - Research Site, Gandia, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Valladolid, Valladolid
  - Research Site, Bilbao, Vizcaya
  - Research Site, Getxo, Vizcaya
  - Research Site, Zalla, Vizcaya
  - Research Site, Benavente, Zamora
  - Research Site, Zaragoza, Zaragoza
  - Research Site, Barcelona